CLINICAL TRIAL: NCT05409352
Title: Effects of Self-administered Acupressure Versus Aerobic Exercise for Treating Cancer-related Fatigue in Cancer Patients Undergoing Chemotherapy: A Randomized Controlled Equivalence Trial
Brief Title: Self-administered Acupressure to Improve Cancer-related Fatigue Among Cancer Patients Undergoing Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Shuk-Ting, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW21084
Record Dates: First submitted 2022-05-30; First posted 2022-06-08 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Cancer, Breast; Fatigue; Acupressure; Exercise
Keywords: cancer; fatigue; acupressure; exercise; chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomization will be performed using software that allows for replication by an independent randomizer. To aid allocation concealment, permuted blocks of varying sizes will be used. The randomizer will place the assignment results in sealed, sequentially numbered opaque envelopes and keep a secure copy of the randomization codes. Neither the research assistant (RA) conducting recruitment nor the participants will know the group assignments until the envelope is opened. All outcome assessments will be carried out by research staff blinded to allocation. Neither the specialist delivering exercise intervention nor the TCM practitioner delivering acupressure intervention will be told about the study design or involved in outcome assessment. The statistician performing data analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-administered acupressure (Experimental): The entire intervention will last 12 weeks, including a one-on-one, 90-min instructional session at week 1 and a one-hour follow-up visit at week 2, which are conducted by a trained traditional Chinese medicine practitioner. Participants will be instructed to perform self-acupressure on the acupoints according to individualized protocol once a day. Participants will be instructed to maintain self-practice after the intervention.
  Interventions: Behavioral: Self-administered acupressure
- Aerobic exercise (Active Comparator): The 12-week aerobic exercise program consists of a one-on-one, 90-min instructional session at week 1 and a one-hour follow-up visit at week 2, which are conducted by a trained exercise specialist. Participants will be advised to perform aerobic exercise of moderate intensity 3 times per week for 30 minutes each time. Accumulating 90 min of exercise per week through more frequent short bouts (e.g. 10-20 min daily) are allowed during the first week of each chemotherapy cycle due to increased symptom burden. Participants will be instructed to maintain self-practice after the intervention.
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Self-administered acupressure — Participants will receive training of self-acupressure on the 5 standard acupoints by a trained traditional Chinese medicine (TCM) practitioner, have return-demonstration, be assessed by the practitioner with the use of a competency checklist, and be instructed to perform self-acupressure on the standard acupoints once a day. A follow-up visit will be conducted to reinforce learning, in which participants will demonstrate the acupressure technique while the practitioner observes and provides feedback, including suggestions for technique adjustments if necessary. The practitioner will recommend 2 additional acupoints from the list of optional acupoints based on the patients' sensitivity to acupoint stimulation and preference. Daily duration of self-practice will range from 8-10 minutes depending on the semi-individualized protocol (5 standard + 2 optional acupoints).
  Arms: Self-administered acupressure
Behavioral: Aerobic exercise — Participants will receive verbal and written information from a trained exercise specialist about the specific advice of the desired exercise frequency (3x/week), duration (30 min each time), and intensity (moderate determined by rating of 12 to 14 on the Borg Rating of Perceived Exertion scale). The exercise specialist will demonstrate how to perform walking at moderate intensity indoors and outdoors, followed by return-demonstration of the patient. Education on safety precautions and walk schedule planning will be provided. Competency check will be performed to assess participants' ability to self-monitor and self-regular exercise intensity using Borg Scale. One week after the start of the program, the exercise specialist will conduct a 1-hour follow-up visit to supervise the patient's walking session and assess whether there is any additional advice needed.
  Arms: Aerobic exercise

SUMMARY:
The primary aim of the study is to determine whether self-administered acupressure has effects equivalent to aerobic exercise on CRF in cancer patients undergoing chemotherapy. Secondary outcomes include sleep disturbance (self-reported and objective), activity levels (self-reported and objective), quality of life (QoL), cognitive impairment, return to work, chemotherapy completion, and adherence to the intervention. This will be a prospective, assessor-blind, parallel group randomized controlled trial (RCT) that will strictly follow the CONSORT guidelines. A total of 138 patients aged 18 or above with a diagnosis of breast cancer scheduled to commence their first cycle of outpatient adjuvant chemotherapy will be recruited and randomized into self-administered acupressure and aerobic exercise groups. The hypothesis of this study is self-administered acupressure and aerobic exercise demonstrate equivalent effects on CRF. The acupressure arm comprises of a one-on-one, 90-min instructional session and a 1-hour follow-up visit by a trained Traditional Chinese Medicine (TCM) practitioner, and self-practice for 12 weeks. The exercise arm consists of a one-on-one, 90-min instructional session and a 1-hour follow-up visit by a trained exercise specialist, and self-practice for 12 weeks. Participants will be instructed to maintain self-practice after the intervention. Intention-to-treat analysis will be performed.

DETAILED DESCRIPTION:
Cancer-related fatigue (CRF) is recognized as the most frequently reported and distressing symptom among cancer patients. CRF is particularly prevalent in patients undergoing chemotherapy, reported to affect 82-100% of such patients, which in some cases may lead to treatment interruption or discontinuation. If CRF is left untreated during chemotherapy, patients are more likely to have clinically significant CRF that persists for months and years after the treatment. CRF has pervasive impact on a patient's mood, ability to perform daily activities, social relationships, and quality of life (QoL). It also imposes significant financial burden by limiting a patient's ability to work. CRF has been shown to be a risk factor of cancer recurrence and shortened survival. In view of its high prevalence and negative impact, combined with growing survival rates, CRF can be considered as a major public health concern.

Aerobic exercise is the most recommended non-pharmacological strategy for CRF, but it has practical limitations due to a number of barriers to exercise during cancer treatment. Self-administered acupressure is emerging as a promising new strategy for reducing CRF in post-treatment disease-free cancer survivors, but has not been tested rigorously among cancer patients receiving chemotherapy. Both exercise and acupressure are inexpensive and safe self-management strategies that can alleviate CRF and co-occurring cancer symptoms, but as acupressure demands less energy, it may thus be acceptable for a wider range of patients undergoing chemotherapy and experiencing CRF. While previous RCTs on acupressure have focused on post-treatment cancer patients, studies targeting patients undergoing cancer treatment are scarce. A rigorously designed RCT of self-administered acupressure among patients receiving chemotherapy is warranted. To date, no study has examined the equivalence of self-administered acupressure and exercise for reducing CRF. Knowledge of the equivalence of aerobic exercise and acupressure for relieving CRF has important clinical implications that could allow practitioners to target recommendations on the basis of patient preference for a particular type of self-care management.

The primary aim of this study is to determine whether self-administered acupressure has effects equivalent to aerobic exercise on CRF in cancer patients undergoing chemotherapy. The hypothesis of this study is self-administered acupressure and aerobic exercise demonstrate equivalent effects on CRF. Secondary outcomes include sleep disturbance (self-reported and objective), activity levels (self-reported and objective), QoL, cognitive impairment, return to work, chemotherapy completion, and adherence to the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 or above
2. with a diagnosis of breast cancer
3. scheduled to commence their first cycle of outpatient adjuvant chemotherapy
4. have an Eastern Cooperative Oncology Group performance status of 0 or 1
5. screened as no contraindications for exercise based on a pre-exercise safety assessment (including aspects of blood results, cardiorespiratory signs and symptoms, metastasis, and variations in cognitive functions)
6. written informed consent

Exclusion Criteria:

1. have received/self-administered acupressure or acupuncture in the previous 3 months
2. have engaged in >90 min of moderate intensity aerobic exercise per week in the previous 3 months
3. are pregnant or lactating
4. have any injury or ulcers around the acupoints
5. unable to communicate in Cantonese, Mandarin, or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Fatigue levels | post-intervention (the week after the 12-week intervention)
  The Brief Fatigue Inventory (BFI, 9 items) will be used to assess fatigue levels. The first 3 items (fatigue severity subscale) ask patients to describe their current, usual, and worst fatigue in the past 24 hours. The next 6 items (interference subscale) ask the extent to which fatigue interferes with various aspects of life. The mean scores of the 9 items can be categorized as mild (1-3), moderate (4-6), and severe (7-10).
Fatigue levels | one month after the end of all chemotherapy cycles
  The Brief Fatigue Inventory (BFI, 9 items) will be used to assess fatigue levels. The first 3 items (fatigue severity subscale) ask patients to describe their current, usual, and worst fatigue in the past 24 hours. The next 6 items (interference subscale) ask the extent to which fatigue interferes with various aspects of life. The mean scores of the 9 items can be categorized as mild (1-3), moderate (4-6), and severe (7-10).

SECONDARY OUTCOMES:
Self-reported sleep quality | post-intervention (the week after the 12-week intervention), one month after the end of all chemotherapy cycles
  The Pittsburgh Sleep Quality Index (PSQI, 19 items) will be used to assess self-reported sleep quality. Seven component scores are formed: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The scores are summed to produce a global score (0 to 21), with higher scores denoting poorer sleep quality.
Health-related quality of life (QoL) | post-intervention (the week after the 12-week intervention), one month after the end of all chemotherapy cycles
  The Functional Assessment of Cancer Therapy-Breast (FACT-B) will be used to assess health-related QoL. It has 5 domains: physical, emotional, social/family, and functional well-being. The higher the total scores, the higher levels of QoL.
Self-reported activity levels | post-intervention (the week after the 12-week intervention), one month after the end of all chemotherapy cycles
  Self-reported activity levels will be measured by the 7-item International Physical Activity Questionnaire short form (IPAQ-SF). Participants will recall types of intensity of physical activity (for estimating total physical activity in metabolic equivalent task-min/week) and sitting time in the last 7 days.
Return to work | one month after the end of all chemotherapy cycles
  Return to work will be calculated as the percentage of work resumption among those in paid employment at the time of diagnosis and absent from work before the start of treatment.
Chemotherapy completion | one month after the end of all chemotherapy cycles
  Chemotherapy completion will be calculated as the percentage of patients who would complete chemotherapy without dose adjustments.
Objective measure of sleep quality and activity levels | post-intervention (the week after the 12-week intervention), one month after the end of all chemotherapy cycles
  Actigraphy will serve as an objective measure of sleep quality and activity levels. The ActiGraph, a non-invasive, wristwatch-sized device, is a widely used, valid, and reliable measure of activity and sleep. Patients will be asked to wear it for three separate 72-hour periods at study entry, post-intervention, one month after the end of all chemotherapy cycles. The parameters of the activity-rest and sleep-wake patterns (e.g., step count, total sleep time, sleep efficiency) will be analyzed by the accompanying software. Participants will record daily activities, bedtimes, and rising times when wearing the device in the diary.
Adherence | post-intervention (the week after the 12-week intervention), one month after the end of all chemotherapy cycles
  Adherence from study entry to post-intervention and from post-intervention to one month after the end of all chemotherapy cycles will be calculated based on the exercise/acupressure diary. Those who have completed ≥ 75% of prescription will be regarded as adherers.
Cognitive impairment | post-intervention (the week after the 12-week intervention), one month after the end of all chemotherapy cycles
  Cognitive impairment will be assessed using the Montreal Cognitive Assessment (MoCA) 5-min and the cognitive functioning subscale of European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30).

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on reasonable request as decided by the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 3 years after the manuscript on main findings is published.